CLINICAL TRIAL: NCT00567255
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study Comparing the Safety and Efficacy of Naltrexone Sustained Release (SR)/Bupropion Sustained Release (SR) and Placebo in Obese Subjects
Brief Title: A Safety and Efficacy Study of Naltrexone SR/Bupropion SR in Overweight and Obese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NB-303; COR-II (Other: Orexigen Therapeutics, Inc.)
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Obesity; Overweight
Keywords: Obesity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NB32 (Experimental): Naltrexone SR 32 mg/bupropion SR 360 mg/day with ancillary therapy
  Interventions: Drug: Naltrexone SR 32 mg/bupropion SR 360 mg/day; Behavioral: Ancillary therapy
- Placebo (Placebo Comparator): Placebo with ancillary therapy
  Interventions: Drug: Placebo; Behavioral: Ancillary therapy

INTERVENTIONS:
Drug: Naltrexone SR 32 mg/bupropion SR 360 mg/day
  Other Names: NB32
  Arms: NB32
Drug: Placebo
  Arms: Placebo
Behavioral: Ancillary therapy — Ancillary therapy consisting of diet instruction, advice on behavior modification, and exercise counseling

SUMMARY:
The purpose of this study is to determine whether the combination of naltrexone SR and bupropion SR is safe and effective in the treatment of obesity.

DETAILED DESCRIPTION:
Two Phase II clinical trials demonstrated that a combination of bupropion SR and naltrexone is associated with greater weight loss than naltrexone alone, bupropion SR alone or placebo in subjects with uncomplicated obesity. The current study investigated the safety and efficacy of the combination of naltrexone SR and bupropion SR compared to placebo in obese subjects with uncomplicated obesity and in those with overweight/obesity and hypertension and/or dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 18 to 65 years (inclusive)
* Body mass index (weight [kg]/height [m²]) ≥30 and ≤45 kg/m² for subjects with uncomplicated obesity, and BMI of ≥27 and ≤45 kg/m² for subjects with obesity with controlled hypertension and/or dyslipidemia
* Normotensive (systolic ≤140 mm Hg and diastolic ≤90 mm Hg). Anti-hypertensive medications were allowed with the exception of alpha-adrenergic blockers and clonidine. Medical regimen was to be stable for at least 6 weeks prior to randomization.
* Medications for the treatment of dyslipidemia were allowed as long as the medical regimen had been stable for at least 6 weeks prior to randomization.
* Free of opioid medication for 7 days prior to randomization
* No clinically significant abnormality of serum albumin, blood urea nitrogen (BUN), creatinine, bilirubin, sodium, potassium, chloride, calcium or phosphorus
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 2.5 times upper limit of normal (ULN)
* No clinically significant abnormality of hematocrit, white blood cell (WBC) count, WBC differential, or platelets
* Fasting glucose <126 mg/dL and not receiving hypoglycemic agents and fasting triglycerides level <400 mg/dL
* No clinically significant abnormality on urinalysis
* Thyroid stimulating hormone (TSH) within normal limits or normal triiodothyronine (T3), if TSH was below normal limits
* Female subjects of childbearing potential had a negative serum pregnancy test
* Negative urine drug screen (UDS)
* An IDS-SR score <2 on individual items: 5 (sadness), 6 (irritability), 7 (anxiety/tension), and 18 (suicidality) and an IDS-SR total score <30
* Female subjects of childbearing potential were non-lactating and agreed to continue to use effective contraception throughout the study and 30 days after discontinuation of study drug
* Able to comply with all required study procedures and schedule
* Able to speak and read English
* Provided written informed consent

Exclusion Criteria:

* Obesity of known endocrine origin (e.g., untreated hypothyroidism, Cushing's syndrome)
* Serious medical condition (including but not limited to renal or hepatic insufficiency; Class III or IV congestive heart failure, history of angina pectoris, myocardial infarction, claudication, or acute limb ischemia within the previous 6 months; lifetime history of stroke)
* History of malignancy within the previous 5 years, with exception of non-melanoma skin cancer or surgically cured cervical cancer
* Lifetime history of serious psychiatric illness, including lifetime history of bipolar disorder, schizophrenia or other psychosis, bulimia, or anorexia nervosa
* Current serious psychiatric illness including severe personality disorder (e.g., borderline or antisocial), current severe major depressive disorder, recent (previous 6 months) suicide attempt, current active suicidal ideation or recent hospitalization due to psychiatric illness
* Response to the bipolar disorder questions that indicated the presence of bipolar disorder
* Required medications for the treatment of a psychiatric disorder (with the exception of short-term insomnia) within the previous 6 months prior to randomization
* History of drug or alcohol abuse or dependence (with the exception of nicotine dependence) within 1 year prior to study initiation
* Type I or Type II diabetes mellitus
* Screening ECG with a corrected QT (QTc) interval (using Bazett's formula >450 millisecond (msec) [males] and >470 msec [females]) or the presence of any clinically significant cardiac abnormalities, including but not limited to patterns consistent with myocardial ischemia, electrolyte abnormalities, or atrial or ventricular dysrhythmia or significant conduction abnormalities
* Received excluded concomitant medications: any psychotropic agents (including antipsychotic, antidepressant, anxiolytic, mood stabilizer or anticonvulsant agents or agents for the treatment of attention deficit disorder) with the exception of low-dose benzodiazepine or hypnotic agents for the treatment of insomnia (up to 2 mg lorazepam/day or equivalent dose of a benzodiazepine or hypnotic agent); any anorectic or weight loss agents; any over the-counter dietary supplements or herbs with psychoactive, appetite or weight effects; alpha-adrenergic blockers; dopamine agonists; clonidine; coumadin; theophylline; cimetidine; oral corticosteroids; cholestyramine; cholestypol; Depo-Provera®; smoking cessation agents; use of opioid or opioid-like analgesics, including analgesics and antitussives
* History of surgical or device (e.g., gastric banding) intervention for obesity
* History of seizures of any etiology, or of predisposition to seizures (e.g., history of cerebrovascular accident, head trauma with ≥5 minutes loss of consciousness, concussion symptoms lasting ≥15 minutes, brain surgery, skull fracture, subdural hematoma, or febrile seizures)
* History of treatment with bupropion or naltrexone within the preceding 12 months
* History of hypersensitivity or intolerance to bupropion or naltrexone
* Initiation or discontinuation of tobacco products including inhaled tobacco (e.g., cigarettes, cigars, pipes, etc), chewing tobacco or snuff within 3 months prior to randomization or planned during study participation. Use of nicotine replacement products (e.g., nicotine gum, patch, etc) during study participation was not allowed
* Used drugs, herbs, or dietary supplements believed to significantly affect body weight or participated in a weight loss management program within one month prior to randomization
* Loss or gained >4.0 kilograms within the previous 3 months prior to randomization
* Females who were pregnant or breast-feeding or planning to become pregnant during the study period or within 30 days of discontinuing study drug
* Planned surgical procedure that could impact the conduct of the study
* Received any investigational drug or used an experimental device or procedure within the previous 30 days
* Participated in any previous clinical trial conducted by Orexigen
* Had any condition that in the opinion of the investigator made the subject unsuitable for inclusion into the study
* Investigators, study personnel, sponsor representatives and their immediate families

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1496 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Lovelace Scientific Resources, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - HealthStar Research, Hot Springs, Arkansas
  - Northern California Research, Carmichael, California
  - Sierra Medical Research, Fresno, California
  - Pharmacology Research Institute, Newport Beach, California
  - Center for Human Nutrition University of Colorado Health Sciences Center, Denver, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Suncoast Clinical Research, Palm Harbor, Florida
  - Comprehensive NeuroScience, Inc, Atlanta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Trover Center for Clinical Studies, Madisonville, Kentucky
  - Nutrition and Weight Mangement Center Boston Medical Center, Boston, Massachusetts
  - Milford Emergency Associates, Inc, Milford, Massachusetts
  - Summit Research Network, Inc., Okemos, Michigan
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - Mercy Health Research, St Louis, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Endocrinology & Diabetes Consultants, Dover, New Hampshire
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Central New York Clinical Research, Manlius, New York
  - Comprehensive Weight Control Program, New York, New York
  - Behavioral Medical Research, Staten Island, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Patient Priority, Cincinnati, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - The Portland Clinic, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mountain View Clinical Research, Greer, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - The Cooper Institute, Dallas, Texas
  - Summit Research Network, Inc., Seattle, Washington

REFERENCES:
- [Result] Apovian CM, Aronne L, Rubino D, Still C, Wyatt H, Burns C, Kim D, Dunayevich E; COR-II Study Group. A randomized, phase 3 trial of naltrexone SR/bupropion SR on weight and obesity-related risk factors (COR-II). Obesity (Silver Spring). 2013 May;21(5):935-43. doi: 10.1002/oby.20309. PMID 23408728

RESULTS

PARTICIPANT FLOW:
Groups:
- NB32: Naltrexone SR 32 mg/bupropion SR 360 mg/day
- Placebo: Placebo
Period: Overall Study
Arm/Group | NB32 | Placebo
Started | 1001 | 495
Completed | 538 | 267
Not Completed | 463 | 228
Not completed — Adverse Event | 241 | 68
Not completed — Lost to Follow-up | 77 | 48
Not completed — Withdrawal by Subject | 75 | 56
Not completed — Lack of Efficacy | 19 | 33
Not completed — Protocol Violation | 20 | 8
Not completed — Pregnancy | 6 | 0
Not completed — Drug noncompliance,moved,other | 25 | 15

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | NB32 | Placebo | Total
Number analyzed (Participants) | 1001 | 495 | 1496
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.27 (11.16) | 44.41 (11.38) | 44.32 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 847 | 420 | 1267
  Male | 154 | 75 | 229
Race/Ethnicity, Customized [Number; unit: participants]
  White | 835 | 414 | 1249
  Black or African American | 133 | 72 | 205
  Asian | 12 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  American Indian or Alaska Native | 10 | 2 | 12
  Other | 8 | 2 | 10
Weight [Mean (Standard Deviation); unit: kg] | 100.3 (16.55) | 99.21 (15.86) | 99.95 (16.33)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.22 (4.45) | 36.09 (4.27) | 36.17 (4.39)

OUTCOME MEASURES:

1. Primary Outcome: Co-primary: Body Weight- Mean Percent Change From Baseline to Week 28
Time Frame: Baseline, 28 weeks
Population: Modified ITT (Full Analysis Set): Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percentage of body weight
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 825 | 456
percentage of body weight | -6.45 (0.20) | -1.89 (0.26)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -4.56, 95% CI [-5.19 to -3.93]

2. Secondary Outcome: Body Weight- Mean Percent Change From Baseline to Week 56
Description: Beginning at Week 28 through Week 44, NB32-treated subjects who failed to achieve or maintain at least 5% body weight loss from baseline were re-randomized (1:1 ratio) to continue NB32 or begin treatment with a higher dose of naltrexone SR - naltrexone SR 48 mg/bupropion SR 360 mg (referred to as NB48) (daily dose of bupropion SR was 360 mg for NB32 and NB48).The analysis of NB32 vs. placebo at Week 56 was completed using a weighted analysis. This analysis was referred to as the weighted LOCF analysis.
  Subjects treated with NB32 who were re-randomized to NB48 were not included. Subjects re-randomized to NB32 were double-weighted and subjects who were not re-randomized were single-weighted. Subjects in the placebo group were single-weighted. The double weighting analysis restored the influence of poor performers at Weeks 28 to 44 in the NB32 group without including any data from the higher dose group (NB48).
Time Frame: Baseline, 56 weeks
Population: Modified ITT: Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percentage of body weight
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 702 | 456
percentage of body weight | -6.40 (0.25) | -1.23 (0.33)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -5.16, 95% CI 2-sided [-5.95 to -4.38]

3. Primary Outcome: Co-primary: Body Weight- Proportion of Subjects With ≥5% Decrease From Baseline to Week 28
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 825 | 456
percentage of participants | 55.64 [52.25 to 59.03] | 17.54 [14.05 to 21.03]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.61, 95% CI [4.95 to 8.84]

4. Secondary Outcome: Body Weight- Proportion of Subjects With ≥5% Decrease From Baseline to Week 56
Description: as for outcome 2
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 702 | 456
percentage of participants | 50.48 [46.90 to 54.07] | 17.11 [13.46 to 20.75]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.50, 95% CI 2-sided [4.05 to 7.47]

5. Secondary Outcome: Body Weight- Proportion of Subjects With ≥10% Decrease From Baseline to Week 28
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 825 | 456
percentage of participants | 27.27 [24.23 to 30.31] | 7.02 [4.67 to 9.36]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.36, 95% CI 2-sided [3.60 to 7.98]

6. Secondary Outcome: Change in Waist Circumference
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 622 | 315
cm | -6.16 (0.28) | -2.74 (0.38)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.43, 95% CI 2-sided [-4.33 to -2.53]

7. Secondary Outcome: Change in Fasting HDL Cholesterol Levels
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 625 | 308
mg/dL | 1.19 (0.30) | -1.40 (0.42)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 2.59, 95% CI 2-sided [1.61 to 3.57]

8. Secondary Outcome: Change in Fasting Triglycerides Levels, Using Log-transformed Data
Time Frame: Baseline, 28 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 625 | 308
percent change | -7.32 [-9.80 to -4.76] | -1.36 [-5.02 to 2.43]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Net) = -5.96

9. Secondary Outcome: Change in IWQOL-Lite Total Scores
Description: IWQOL-Lite= Impact of Weight on Quality of Life-Lite Questionnaire Total score is based on a scale from 0 to 100, with 0 representing the poorest and 100 the best quality of life and where a score of 71-79 indicates moderate impairment
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 628 | 317
units on a scale | 9.94 (0.41) | 6.17 (0.56)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 3.77, 95% CI 2-sided [2.46 to 5.09]

10. Secondary Outcome: Change in High-sensitivity C Reactive Protein (Hs-CRP) Levels, Using Log-transformed Data
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 607 | 304
percent change | -9.38 [-14.78 to -3.63] | -1.14 [-9.11 to 7.52]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.091, ANCOVA; Mean Difference (Net) = -8.24

11. Secondary Outcome: Change in Fasting Insulin Levels, Using Log-transformed Data
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 589 | 286
percent change | -14.14 [-17.86 to -10.24] | -0.50 [-6.49 to 5.88]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -13.64

12. Secondary Outcome: Change in Fasting Blood Glucose Levels
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 628 | 310
mg/dL | -2.11 (0.38) | -1.73 (0.52)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.38, 95% CI 2-sided [-1.60 to 0.85]

13. Secondary Outcome: Change in HOMA-IR Levels, Using Log-transformed Data
Description: HOMA-IR= Homeostasis Model Assessment-Insulin Resistance
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 580 | 278
percent change | -16.44 [-20.37 to -12.31] | -4.15 [-10.43 to 2.57]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -12.29

14. Secondary Outcome: Change in Question 19 From 21-Item COE (Control of Eating) Questionnaire
Description: Question 19: Generally, how difficult has it been to control your eating? Scoring: 0=not at all difficult; 100=extremely difficult
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 731 | 409
units on a scale | -18.32 (0.85) | -11.09 (1.12)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -7.23, 95% CI 2-sided [-9.92 to -4.54]

15. Secondary Outcome: Change in Fasting LDL Cholesterol Levels
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 620 | 308
mg/dL | -4.36 (0.90) | 0.00 (1.25)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -4.36, 95% CI 2-sided [-7.29 to -1.44]

16. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 824 | 456
mm Hg | -0.93 (0.31) | -1.23 (0.42)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.30, 95% CI 2-sided [-0.70 to 1.30]

17. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 824 | 456
mm Hg | 0.20 (0.22) | -0.67 (0.30)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.87, 95% CI 2-sided [0.16 to 1.58]

18. Secondary Outcome: Change in IDS-SR Total Score
Description: IDS-SR= Inventory of Depressive Symptoms-Subject Rated IDS-SR total score is based on 30 items. The total score can range from 0-84, with 0 being no depressive symptoms and 84 being very severe depressive symptoms. A total score ≤ 13 indicates no depression.
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 825 | 455
units on a scale | -0.23 (0.17) | -0.28 (0.23)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.49 to 0.60]

19. Secondary Outcome: Change in Food Craving Inventory Sweets Subscale Score
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The sweets subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 753 | 418
units on a scale | -3.20 (0.17) | -3.18 (0.22)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.56 to 0.52]

20. Secondary Outcome: Change in Food Craving Inventory Carbohydrates Subscale Score
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The carbohydrates subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 28 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 754 | 418
units on a scale | -2.68 (0.16) | -2.20 (0.21)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.98 to 0.02]

ADVERSE EVENTS:
Time Frame: Baseline, 56 weeks
Description: The safety analysis set includes all randomized subjects who took study drug and were assessed by investigator after their first dose, whether or not they discontinue the study. Treatment-emergent adverse events were defined as events that started or worsened in the double-blind treatment phase after the first dose and before 7 days post last dose.
Groups:
- NB32/48: Naltrexone SR 32 mg/bupropion SR 360 mg/day or naltrexone SR 48 mg/bupropion SR 360 mg/day
  Beginning at Week 28 through Week 44, NB32-treated subjects who failed to achieve or maintain at least 5% body weight loss from baseline were re-randomized (1:1 ratio) to continue NB32 or begin treatment with a higher dose of naltrexone SR - naltrexone SR 48 mg/bupropion SR 360 mg (referred to as NB48) (daily dose of bupropion SR was 360 mg for NB32 and NB48).
  NB32/48 group includes all participants in the safety analysis set randomized to NB32 at baseline, regardless of re-randomization status.
Arm/Group | NB32/48 | Placebo
Serious Adverse Events (participants affected / at risk) | 21/992 | 7/492
Other Adverse Events (participants affected / at risk) | 671/992 | 244/492
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32/48 (N=992) | Placebo (N=492)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32/48 (N=992) | Placebo (N=492)
Constipation (Gastrointestinal disorders) | 189 (199) | 35 (36)
Diarrhoea (Gastrointestinal disorders) | 55 (57) | 18 (21)
Dry mouth (Gastrointestinal disorders) | 90 (91) | 13 (13)
Nausea (Gastrointestinal disorders) | 290 (329) | 34 (41)
Vomiting (Gastrointestinal disorders) | 84 (95) | 10 (10)
Bronchitis (Infections and infestations) | 14 (14) | 25 (26)
Nasopharyngitis (Infections and infestations) | 82 (93) | 40 (45)
Sinusitis (Infections and infestations) | 51 (63) | 35 (41)
Upper respiratory tract infection (Infections and infestations) | 86 (98) | 55 (70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (42) | 28 (30)
Dizziness (Nervous system disorders) | 68 (76) | 17 (19)
Headache (Nervous system disorders) | 174 (197) | 43 (47)
Insomnia (Psychiatric disorders) | 97 (106) | 33 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 18 months after conclusion of the study at all study centers, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 60 days to review and comment on the proposed publication. The review period may be extended by an additional 30 days upon request. Sponsor may delay publication for up to an additional 6 month period to file for patent protection.